CLINICAL TRIAL: NCT05660239
Title: Epilepsy in Uganda: Clinical Characterization and Co-morbidities, Their Relation to Stigma Among Adolescents and Impact of a Community-based Engagement Program
Brief Title: Impact of a Community Based Engagement Program Focused on Adolescents With Epilepsy
Acronym: AWE-Change
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R01HD106277-01 (NIH); R01HD106277 (NIH)
Record Dates: First submitted 2022-12-07; First posted 2022-12-21 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Study participants together with the relevant community stakeholders will co-design feasible communication and activity-based change projects that are based on both cultural and scientific norms, to reduce epilepsy stigma in the community Researchers will then compare the Quality of Life, Attitudes and Beliefs about Living with Epilepsy scores and the Kilifi Stigma Scale scores, pre and post the implementation of the community change projects in two parishes (urban and rural) to see if there is improvement in these assessments scores.
Who Masked: Outcomes Assessor
Masking Description: Study participants and researchers both know which community change intervention they are receiving or implementing respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wakiso district-Urban Parish (Other): Study participants together with the relevant community stakeholders will co-design feasible communication and activity-based change projects that are based on both cultural and scientific norms, to reduce epilepsy stigma in the community.
  Researchers will then compare the Quality of Life, Attitudes and Beliefs about Living with Epilepsy scores and the Kilifi Stigma Scale scores following the implementation of the community change projects in an urban parish to see if there is improvement in these assessments scores.
  Interventions: Other: Community Intervention
- Wakiso district-Rural Parish (Other): Study participants together with the relevant community stakeholders will co-design feasible communication and activity-based change projects that are based on both cultural and scientific norms, to reduce epilepsy stigma in the community.
  Researchers will then compare the Quality of Life, Attitudes and Beliefs about Living with Epilepsy scores and the Kilifi Stigma Scale scores following the implementation of the community change projects in a rural parish to see if there is improvement in these assessments scores.
  Interventions: Other: Community Intervention

INTERVENTIONS:
Other: Community Intervention — To evaluate the impact of a community intervention in reducing epilepsy stigma in adolescents.

SUMMARY:
The goal of this community based observation study is to co-create solutions that empower people to make informed decisions about epilepsy, reduce stigma, and promote community health among the adolescent population living with epilepsy in Uganda.

The main objectives of the study are to:

Goal 1: Co-create a unique patient-community engagement program (CEP) to reduce stigma on epilepsy among adolescents and their caregivers in Uganda based on understanding of the illness.

Goal 2: Evaluate the impact of this CEP to reduce stigma on epilepsy among adolescents and their caregivers in Uganda, based on understanding of the illness.

Study participants together with the relevant community stakeholders will co-design feasible communication and activity-based change projects that are based on both cultural and scientific norms, to reduce epilepsy stigma in the community Researchers will then compare the Quality of Life, Attitudes and Beliefs about Living with Epilepsy scores (as a surrogate of stigmatizing beliefs and practices among community members) and the Kilifi Stigma Scale scores in two parishes (urban and rural) to see if there is improvement in these assessments scores following the implementation of the community change projects.

DETAILED DESCRIPTION:
Study Site:

The study will be conducted in Wakiso District which lies in the Central region of Uganda with a target adolescent group (ages 10-18) comprising ~22% of the population. Wakiso District has the largest population density and a 7% growth rate. Our previous epilepsy prevalence work also showed it had the highest number of adolescents with epilepsy (AWE). Wakiso also offers the advantage of having both rural communities similar to those in more remote areas of the country, as well as rapidly expanding urban communities as seen in other urban centers like Kampala city, the capital.

Selecting the communities for intervention:

Two Wakiso district divisions will be randomly selected from enumerated divisions. Within these, parishes will be enumerated and divided into urban and rural parishes, from which one rural and one urban will be randomly selected. The investigators will then list the villages within each selected parish and randomly select two adjacent villages per parish. Using Objective 1 records, the investigators will contact AWE (ages 10-18) and their caregivers in these villages for invitation to the CEP, and the investigators will repeat this step as needed until the required number is obtained.

Study Implementation:

Step 1: a) Evaluate tacit knowledge and values of community stakeholders. Methods: focus groups discussions (FGDs), in depth interviews, and social media discussions with community leaders, clergy, traditional healers, teachers, and any people who are agents of progression and change. For the in depth interviews the investigators plan to engage 20-40 stakeholders, while for the focus group discussions about 10-20, the stakeholders will be categorized according to their gender and respective age groups in groups of 6-8 individuals per FGD until data saturation is achieved. b) Obtain baseline Attitudes and Beliefs about Living with Epilepsy (ABLE) scale scores. c) Select the stigma reduction implementation team (SRIT)- this will involve a smaller group of participants, called the SRIT, composed of patient champions (AWE and/or their caregivers; n=5-10), community champions (n=5-10), and members of the research team will convene to plan communication and activity-based change solutions that are based on both cultural and scientific norms of all stakeholders. This participatory approach to problem solving is a proven method to optimize change management.

Step 2: Enhance and refine epilepsy knowledge within the SRIT by cultivating shared culturally and scientifically informed perspectives. With identification of key areas of concern regarding epilepsy stigma, communities and other stakeholders of epilepsy for example Epilepsy Support Association, Uganda (ESAU) or Purple Bench Initiative will also be engaged in various dialogue forms to identify solutions to the issues identified.

Step 3: Co-create strategies for paradigm change; select most promising projects. These culturally and scientifically informed solutions may involve several communication venues, such as packaging messages in poems/songs/drama skits to be delivered through technology-based approaches such as social media, use of social network sites, text messaging, podcasts, blogs, and/or YouTube videos. The SRIT will analyze the merit of all proposed solutions and rank them according to potential for meeting the goals of the engagement within resource guidelines. This ensures investment in the innovative problem-solving practices as utilizing self-management and positive reinforcement within the impacted community. Four full prototypes will be co-created and co-designed to reduce stigma. Two knowledge cycles will inform the development and refinement of the projects to facilitate engagement and new norms Step 4: Implement unique SRIT change projects in the community, monitor project progress for adjustment.

After Cycle 1, progress is jointly evaluated from all stakeholder perspectives, projects are refined or replaced, and Cycle 2 is initiated to impact social change through re-engaging the broad community.

ELIGIBILITY:
Inclusion Criteria:

Adolescent with epilepsy residing in Wakiso district

* Between the ages 10-18 years
* A resident of Wakiso district, Uganda for the previous six months
* Confirmed diagnosis for epilepsy as per the International League Against Epilepsy definition
* Provide written assent to participation in the study
* With a caregiver willing to provide written informed consent as well as detailed history regarding them.
* Willing to participate in all the required program activities with his/her caregiver

Exclusion Criteria:

Adolescent with epilepsy residing in Wakiso district who

* Does not have the time or interest to participate in the community engagement program
* Has had exposure to a similar previous community engagement program
* Is unable to fully understand what is required of him/her in the study and engage consistently throughout the whole community engagement program

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Attitudes and Beliefs about Living with Epilepsy (ABLE) scores among the community stigma reduction implementation team. | two years
  Change in knowledge, attitude and beliefs regarding epilepsy among the community stigma reduction implementation team. Attitudes and Beliefs about Living with Epilepsy (ABLE) scale, are scored on a five-point Likert scale (1=no stigma, 5=high stigma)
Attitudes and Beliefs about Living with Epilepsy (ABLE) scores among the non-community stigma reduction implementation team. | two years
  Change in knowledge, attitude and beliefs regarding epilepsy among the non-community stigma reduction implementation team. Attitudes and Beliefs about Living with Epilepsy (ABLE) scale, are scored on a five-point Likert scale (1=no stigma, 5=high stigma).
Kilifi Stigma Scale scores among adolescents with epilepsy | two years
  Change in perceived stigma for the adolescents living with epilepsy. Kilifi Stigma scale has a three-point Likert scoring, (0 = not at all, 1 = sometimes, 2 = always). A total score is calculated by addition of all item scores. The higher the score, the greater the sense of perceived stigma.
Quality of Life for Epilepsy in Adolescents scores | two years
  Change in the quality of life for the adolescents living with epilepsy. Quality of Life(QoL) for Epilepsy in Adolescents scores are on a 5-point Likert scale with: 1 = poor; and 5 = excellent. Ratings are linearly transformed, providing total scores from 0 (low QoL) to 100 (high QoL).

SECONDARY OUTCOMES:
Beck Youth Inventory for depression (BDI-Youth) scores among adolescents with epilepsy | two years
  Change in the depression severity among adolescents with epilepsy.Beck Youth Inventory for depression (BDI-Youth) raw scores are translated into T-scores assigned by age and gender as follows ( 55 or less = average ; 70+ = extremely elevated).
Columbia Suicide Severity Rating Scale (C-SSRS) scores for the adolescents living with epilepsy. | two years
  Change in the suicide severity among adolescents with epilepsy. There are no specified clinical cutoffs for the Columbia-Suicide Severity Rating Scale due to the binary nature (yes/no) of the responses to 10 category items. Composite endpoints based on the categories as follows:
  Suicidal ideation: A "yes" answer at any time during treatment to any one of the five suicidal ideation questions (Categories 1-5) on the Columbia-Suicide Severity Rating Scale.
  Suicidal behavior: A "yes" answer at any time during treatment to any one of the five suicidal behavior questions (Categories 6-10) on the Columbia-Suicide Severity Rating Scale.
  Suicidal ideation or behavior: A "yes" answer at any time during treatment to any one of the ten suicidal ideation and behavior questions (Categories 1-10) on the Columbia-Suicide Severity Rating Scale.